CLINICAL TRIAL: NCT02643615
Title: A Pilot Study to Determine the Efficacy and Safety of Detecting Subtle Visual Changes During Visual Evoked Potential (VEP) Monitoring Using SightSaver ™ Flash Visual Evoked Potential Stimulator in Spine Prone Surgery
Brief Title: Safety and Efficacy of Using SightSaver Visual Evoked Potential (VEP) for VEP Monitoring in Prone Spine Surgery
Acronym: SightSaver
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Sergio Bergese, Principle Investigator, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2014H0208
Record Dates: First submitted 2015-12-11; First posted 2015-12-31 (Estimated); Results first posted 2017-08-01 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Ischemic Optic Neuropathy
Keywords: Visual Evoked Potentials
MeSH Terms: conditions — Optic Neuropathy, Ischemic | interventions — Propofol; Desflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- VEP under TIVA (Experimental): Patients undergoing prone spine surgery will receive an anesthesia regimen using propofol (TIVA) for maintenance
  Interventions: Device: VEP under TIVA; Drug: Propofol
- VEP under balanced anesthesia (Experimental): Patients undergoing prone spine surgery will receive an anesthesia regimen using Desflurane as part of balanced general anesthesia
  Interventions: Device: VEP under balanced anesth.; Drug: Desflurane

INTERVENTIONS:
Device: VEP under TIVA — Propofol will be administered for anesthesia maintenance in patients randomized to the TIVA arm of the study. In order to record the VEPs, standard half-inch sub-dermal needle electrodes will be inserted subcutaneously around the visual area and the SightSaverTM visual stimulator will be placed to monitor VEP during surgery.
  Arms: VEP under TIVA
Device: VEP under balanced anesth. — Balanced general anesthesia with desflurane will be administered for anesthesia maintenance in patients randomized to the balanced general anesthesia arm of the study, In order to record the VEPs, standard half-inch sub-dermal needle electrodes will be inserted subcutaneously around the visual area and the SightSaverTM visual stimulator will be placed to monitor VEP during surgery.
  Arms: VEP under balanced anesthesia
Drug: Propofol — Propofol will be administered for anesthesia maintenance in patients randomized to the TIVA arm of the study. In order to record the VEPs, standard half-inch sub-dermal needle electrodes will be inserted subcutaneously around the visual area and the SightSaverTM visual stimulator will be placed to monitor VEP during surgery.
  Other Names: Diprivan
  Arms: VEP under TIVA
Drug: Desflurane — Balanced general anesthesia with desflurane will be administered for anesthesia maintenance in patients randomized to the balanced general anesthesia arm of the study, In order to record the VEPs, standard half-inch sub-dermal needle electrodes will be inserted subcutaneously around the visual area and the SightSaverTM visual stimulator will be placed to monitor VEP during surgery.
  Other Names: Suprane
  Arms: VEP under balanced anesthesia

SUMMARY:
Post-operative visual loss (POVL) following non-ocular surgical procedures is an infrequent but severe complication. Little is understood about this complication, but most cases seem to result from loss of blood flow to the optic nerve. This is a pilot, single center, prospective, randomized, two-arm study involving 20 subjects at The Ohio State University Wexner Medical Center who are scheduled to undergo spine surgery that requires prone position and at least two hours of general anesthesia or total intravenous anesthesia (TIVA) and intraoperative neurophysiological monitoring. Patients will be randomized to either general anesthesia or TIVA, and wear the SightSaver device to monitor visual evoked potentials (VEPs) during surgery in order to detect possible changes in optic nerve function that may lead to POVL. We hypothesize that this new, flexible, disposable device will yield better results and more patient satisfaction than devices currently used for visual monitoring during prone spine surgeries.

DETAILED DESCRIPTION:
The exact mechanism underlying POVL is poorly understood, but nearly all cases seem to involve ischemic optic neuropathy (ION). Posterior ION is more commonly the result of spinal procedures. The spine surgery associated risk factors include: prone position, Trendelenburg positioning, blood loss, prolonged procedure, use of vasoconstriction agents to correct blood pressure, direct ocular compression, and hypotension [1,2]. Given the fact that the suspected mechanism is a gradual infarction of the optic nerve, POVL could theoretically be prevented based on early detection of reversible optic nerve dysfunction. Visual evoked potentials (VEP) are a highly sensitive method for detecting optic nerve dysfunction, including ischemia.

During intraoperative neurophysiological monitoring (IONM), an emitted light passes through the lens, reaching the retina and causing hyperpolarization. The signal generated by the retina in response to a flash of light is known as the electroretinogram (ERG). This response may be recorded using conventional neurophysiological equipment and reflects overall retinal function. The VEP peaks are generated during the passage of electrical signal from the retina via the optic pathways to the primary visual cortex, and can also be registered during IONM. Measurements of VEP peaks under anesthesia can vary depending on type of anesthetic regimen, some producing more interference with the electrical impulses than others.

The problems encountered during VEP monitoring are numerous: a reusable device must be cleaned in between patients, tightly fitting goggles pose a risk of damaging the eyes, goggles may fall off or move intraoperatively and be difficult to reposition once the procedure is underway. Also, the light emitting diodes tend to be too weak to produce an adequate stimulus. This pilot study presents a new different approach from current methods. The SightSaverTM visual stimulator design consists of the following key advantages over the current technologies: hygienically superior to re-usable goggles, provides physical protection to the ocular region, use of higher intensity diodes and adhesive foam padding shaped to contours of periocular region.

This pilot, single center, prospective, randomized, two-arm study will involve 20 subjects at The Ohio State University Wexner Medical Center who are scheduled to undergo spine surgery that requires prone position and at least two hours of general anesthesia or TIVA and intraoperative neurophysiological monitoring. Eligible subjects that provide voluntary and written informed consent will be included in the study with a 1:1 randomization ratio of two arms, n=10 patients per each of two anesthesia regimen groups: general anesthesia and TIVA. All patients will wear the SightSaverTM visual stimulator. IONM of VEP with include insertion of half-inch needle electrodes placed just under the skin on either side of the eye, at the top of the forehead and three along the back of the head. Flashes of light, delivered at continuous intervals, will be emitted from diodes mounted in the SightSaverTM visual stimulator. After the baseline VEP is established for the patient, monitoring of VEP will occur at every 30 minutes during surgery. If during the monitoring process, a significant VEP waveform change has occurred, an alert will trigger the surgical staff to check four different parameters: technical issues with goggles, anesthetic changes, significant blood loss or a blood pressure change. Analysis of data collected will be used to evaluate the efficacy of SightSaverTM visual stimulator for intraoperative VEP-based detection of significant visual changes during prone spine surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female older than 18 years of age
* American Society of Anesthesiologists (ASA) status of I to IV and scheduled to undergo elective spinal prone position procedures under general anesthesia or TIVA only with intraoperative neurophysiological monitoring with an expected duration of surgery to be at least 2 hours
* If female, have been surgically sterilized or are postmenopausal; if of child-bearing potential, must have a negative serum pregnancy test the day of surgery
* Ability and willingness to sign informed consent
* Literate in the English language

Exclusion Criteria:

* Prisoner status
* Women who are pregnant or lactating/breast feeding
* Patients with a history of contact allergies to foam and/or plastic devices
* Any condition, which, in the opinion of the investigator, would make the subject ineligible for participation in the study, such as a history of unstable cardiovascular, pulmonary, renal, hepatic, neurologic (seizures), hematologic or endocrine abnormality (hyperthyroidism, unstable Diabetes type I/II)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergio D Bergese, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Enrolled subjects will be assigned a subject identification number and we will not collect any identifiable data

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VEP Under TIVA | VEP Under Balanced Anesthesia
Started | 9 | 11
Completed | 9 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- VEP Under Balanced Anesthesia: Patients undergoing prone spine surgery will receive an anesthesia regimen using Desflurane as part of balanced general anesthesia
  VEP under balanced anesth.: Balanced general anesthesia with desflurane will be administered for anesthesia maintenance in patients randomized to the balanced general anesthesia arm of the study, In order to record the VEPs, standard half-inch sub-dermal needle electrodes will be inserted subcutaneously around the visual area and the SightSaverTM visual stimulator will be placed to monitor VEP during surgery.
  Desflurane: Balanced general anesthesia with desflurane will be administered for anesthesia maintenance in patients randomized to the balanced general anesthesia arm of the study, In order to record the VEPs, standard half-inch sub-dermal needle electrodes will be ins
- Total: Total of all reporting groups
Arm/Group | VEP Under TIVA | VEP Under Balanced Anesthesia | Total
Number analyzed (Participants) | 9 | 11 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 11 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (14.8) | 56.2 (16.1) | 54.5 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 3 | 7 | 10
Region of Enrollment [Number; unit: participants]
  United States | 9 | 11 | 20

OUTCOME MEASURES:

1. Primary Outcome: Efficacy in Detecting Subtle Intraoperative VEP Changes Using SightSaver Visual Stimulator During Spine Prone Surgeries Under Balanced General Anesthesia Versus TIVA.
Description: Number of Participants with Subtle Intraoperative VEP Changes Observed Using SightSaver Visual Stimulator During Spine Prone Surgeries Under Balanced General Anesthesia Versus TIVA
Time Frame: VEP waveforms recorded every 30 minutes during the entire procedure for up to 6 hours.
Measure: Count of Participants; unit: Participants
Arm/Group | VEP Under TIVA | VEP Under Balanced Anesthesia
Number analyzed (Participants) | 9 | 11
Participants | 1 | 1

2. Secondary Outcome: The Difference in VEP Changes in Amplitude Among Both Groups
Description: VEP waveforms were evaluated using either present baseline - reproducible positive-negative-positive complex of substantial amplitude (≥2 µV) that appeared 100-200 ms after pulse stimulus onset; marginal Baseline - low amplitude (<2 µV) reproducible P100 waveform; or absent baseline - no repeatable response present. Any activity of <0.5 µV was not considered a response. Best derivation for each particular patient was used for monitoring electroretinogram (ERG) recording and confirming the stimulation.
Time Frame: Every 30 minutes during surgery for up to 6 hours
Measure: Median (95% Confidence Interval); unit: micorvolts (µV)
Arm/Group | VEP Under TIVA | VEP Under Balanced Anesthesia
Number analyzed (Participants) | 9 | 11
micorvolts (µV) | 0.66 [0.25 to 1.08] | 0.48 [0.06 to 0.90]

3. Secondary Outcome: The Difference in VEP Changes in Amplitude Among Both Groups
Description: The difference in VEP changes in amplitude with a single and double stimuli using the SightSaver visual stimulator under balanced general anesthesia versus TIVA.
Time Frame: every 30 minutes during the entire procedure for up to 6 hours
Measure: Mean (95% Confidence Interval); unit: milliseconds (ms)
Arm/Group | VEP Under TIVA | VEP Under Balanced Anesthesia
Number analyzed (Participants) | 9 | 11
milliseconds (ms) | 14.21 [9.5 to 19.0] | 17.94 [12.8 to 23.0]

4. Secondary Outcome: Safety of Using SightSaver Visual Stimulator During Spine Prone Surgeries Under Balanced General Anesthesia Versus TIVA
Description: Number of participants experiencing adverse events related to the study procedures during prone surgery and 24 hours after surgery under balanced general anesthesia versus TIVA
Time Frame: From start of surgery up to 24 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | VEP Under TIVA | VEP Under Balanced Anesthesia
Number analyzed (Participants) | 9 | 11
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Serious adverse events were recorded during the first 24 hours from anesthesia start time.
Arm/Group | VEP Under TIVA | VEP Under Balanced Anesthesia
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/11
Other Adverse Events (participants affected / at risk) | 0/9 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes